CLINICAL TRIAL: NCT05015582
Title: Randomized Control Trial Assessing Effectiveness of Perioperative Warming Measures in Parturients Undergoing Cesarean Delivery
Brief Title: Perioperative Warming Measures in Cesarean Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Stacy Lynn Norrell, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-21-0011
Record Dates: First submitted 2021-07-22; First posted 2021-08-20 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Hypothermia; Anesthesia; Hypothermia, Newborn; Hypothermia, Sequela
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Treatment (Experimental): Preop: Use of full body forced air warming pre-operative at ambient (32˚C) for at least 30 minutes and fluids from warmed cabinet set at 45˚C
  Intraop: Use of upper body and lower forced air warming intra-operative at 32 and 42˚C respectively and IV fluids with hotline fluid warmer set at 42˚C
  Interventions: Device: Pre op upper body forced air warming (32˚C); Device: Pre op lower body forced air warming (32˚C); Device: Pre op fluids (45˚C); Device: Intra op upper body forced air warming (32˚C); Device: Intra op upper body forced air warming at (32˚C); Device: Intra op upper body forced air warming at (42˚C); Device: Intra op lower body forced air warming at (32˚C); Device: Intra op lower body forced air warming at (42˚C); Device: Intra op fluid (42˚C)
- Control Group (Active Comparator): Preop: Use of full body forced air warming pre-operative at ambient (32˚C) for at least 30 minutes and fluids from warmed cabinet set at 45˚C
  Intraop: Use of upper body forced air warming intra-operative at ambient (32˚C) and IV fluids at room temperature
  Interventions: Device: Pre op upper body forced air warming (32˚C); Device: Pre op lower body forced air warming (32˚C); Device: Pre op fluids (45˚C); Device: Intra op upper body forced air warming (32˚C); Device: Intra op fluids at room temperature; Device: Intra op upper body forced air warming at (32˚C)

INTERVENTIONS:
Device: Pre op upper body forced air warming (32˚C) — Use of upper body forced air warming at ambient (32˚C) for at least 30 minutes
Device: Pre op lower body forced air warming (32˚C) — lower body forced air warming at ambient (32˚C) for at least 30 minutes
Device: Pre op fluids (45˚C) — fluids from warmed cabinet set at 45˚C
Device: Intra op upper body forced air warming (32˚C) — Use of upper body forced air warming intra-operative at ambient (32˚C)
Device: Intra op fluids at room temperature — IV fluids at room temperature
  Arms: Control Group
Device: Intra op upper body forced air warming at (32˚C) — upper body forced air warming intra-operative at ambient (32˚C)
Device: Intra op upper body forced air warming at (42˚C) — upper body forced air warming intra-operative at ambient (42˚C)
  Arms: Treatment
Device: Intra op lower body forced air warming at (32˚C) — Lower body forced air warming intra-operative at ambient (32˚C)
  Arms: Treatment
Device: Intra op lower body forced air warming at (42˚C) — Lower body forced air warming intra-operative at ambient (42˚C)
  Arms: Treatment
Device: Intra op fluid (42˚C) — IV fluids with hotline fluid warmer set at 42˚C
  Arms: Treatment

SUMMARY:
The purpose of this study is to evaluate the best method for keeping patients warm during cesarean deliveries and the effect of temperature change on the patient and baby

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective cesarean section under neuraxial anesthesia
* singleton pregnancy

Exclusion Criteria:

* gestational age of less than 37 week
* emergency cesarean

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in maternal core body temperature | preoperative/beginning of surgery ,postoperative/end of surgery (4 hours after anesthesia)
Number of women with hypothermia | preoperative/beginning of surgery ,postoperative/end of surgery (4 hours after anesthesia)
  Hypothermia is indicated as core temperature < 36 °C
Neonate status as determined by Appearance, Pulse, Grimace, Activity, and Respiration (APGAR) score | 10 minutes after birth
  Five criteria are scored and each one is scored form 0-2 with a total score of 10, a higher score indicating a better outcome.
Neonate status as determined by Umbilical Artery PH | 10 minutes after birth
  determined by lab value
Maternal Coagulopathy | end of surgery (4 hours after anesthesia)
  determined by lab value

SECONDARY OUTCOMES:
Degree of shivering (severity) | on arrival to Post anesthesia Care Unit (PACU) [about 4 hours after anesthesia]
  Degree of shivering is measured from 0(no shivering)-3(total body shivering)
Number of patients that need meperidine | on arrival to PACU [about 4 hours after anesthesia]
Degree of shivering (severity) | after 30 minutes in PACU
  Degree of shivering is measured from 0(no shivering)-3(total body shivering)
Number of patients that need meperidine | after 30 minutes in PACU
Degree of shivering (severity) | after administration of meperidine, if it applies (about 30 minutes in PACU)
  Degree of shivering is measured from 0(no shivering)-3(total body shivering)
Number of patients that show Maternal thermal comfort | end of surgery (4 hours after anesthesia)
  scored form 0-10,a higher number indicating more thermal comfort
Perioperative blood loss | end of surgery (4 hours ater anesthesia)
Hospital Length of Stay | Time of admission to time of discharge (about 72 hours after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Norrell, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No